CLINICAL TRIAL: NCT02615210
Title: Mid-Atlantic Research Group Single-Operator Cholangioscopic Assessment of Biliary Strictures
Acronym: SOCABS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with contracting
Sponsor: Temple University (Other)
Collaborators: Thomas Jefferson University (Other); University of Pennsylvania (Other); University of Pittsburgh Medical Center (Other); Geisinger Clinic (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23154
Record Dates: First submitted 2015-09-22; First posted 2015-11-26 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (No Intervention): Standard of care biopsies with optional SOC-directed biopsy afterwards
- Study (Experimental): SOC-directed biopsies using the SpyGlass System plus standard of care biopsies
  Interventions: Device: SOC-directed biopsies using the SpyGlass System

INTERVENTIONS:
Device: SOC-directed biopsies using the SpyGlass System — The cholangioscopy procedure with the SpyGlass System is performed by a single operator with the SpyScope Access and Delivery Catheter positioned just below the operating channel of the duodenoscope. SpyBite Biopsy Forceps guided by the SpyScope Catheter are introduced and endoscopic-guided biopsy is taken at the level of the stricture. Target lesions will be identified under direct visualization using the SOC system, and 6-8 bites will be performed with the SpyBite forceps. Once SOC-directed biopsies are obtained, the SOC system will be withdrawn into the working channel of the duodenoscope and removed Patient will be contacted monthly to determine if they have undergone any additional procedures and to record potential adverse events.
  Arms: Study

SUMMARY:
The purpose of this study is to determine if cholangioscopically-directed biopsies provide a higher diagnostic yield for malignancy in the setting of indeterminate biliary strictures when compared to standard means of sampling.

DETAILED DESCRIPTION:
Biliary strictures in the absence of a mass are a clinical challenge, as current accepted means of sampling provide suboptimal accuracy. Both biliary brushings for cytology and fluoroscopically-directed biopsies produce highly-variable results. Endoscopic ultrasound with fine-needle aspiration has also been employed with variable results. An additional modality, using a single-operator cholangioscope during endoscopic retrograde cholangiopancreatography (ERCP) to obtain cholangioscopically-directed biopsies offers promise in increasing the yield of sampling. Initial observational studies have shown an improved diagnostic yield, but the technique has not been tested in a randomized, medical effectiveness study to better characterize its actual clinical impact. We aim to compare the technique of biopsy-on-biopsy derived sampling via single-operator cholangioscopy with standard fluoroscopically-directed biopsies and brushings in a pilot study. We also aim to perform a medical effectiveness study on the early use of single-operator cholangioscopically (SOC) in the evaluation of undiagnosed biliary strictures.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Presence of indeterminate biliary strictures with clinical indications for ERCP. Strictures are considered indeterminate when evaluation including cross-sectional imaging is non-diagnostic. Patients who have previously undergone ERCP with sampling will be included, as well as those who have not previously undergone ERCP.
* Strictures located above the intrapancreatic bile duct
* The Subject's physician determines and ERCP is clinically indicated
* Able to provide informed consent

Exclusion Criteria:

* Prior enrollment in the study or another study evaluating biliary strictures
* Presence of extrahepatic malignancy or previously-diagnosed hepatocellular carcinoma
* Pregnancy
* At-risk populations including prisoners and mentally challenged
* Unwilling to provide informed consent
* Medically unfit to undergo ERCP
* History of liver transplant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of malignant diagnoses across hree-sample techniques (Spy bite, forceps biopsy, brushings) | 72 Hours
  Accuracy, sensitivity, and specificity of the three-sample technique (Spy bite, forceps biopsy, brushings) compared to the two-sample technique (forceps biopsy and brushing) in differentiating malignant from benign biliary strictures

SECONDARY OUTCOMES:
Number of patients who receive additional diagnostic studies without receiving a cancer diagnosis | 1 year
  Patients who receive a repeat ERCP with sampling, cross-sectional imaging, EUS-FNA, IR-guided biopsies, laparoscopy
Endoscopic Satisfaction with SOC-directed biopsy | 2 hours
  Endoscopist subjective outcomes using a Likert scale 1-5
  * Ease of obtaining the biopsies
  * Confidence that the biopsy was taken from the target lesion
  * Confidence that an adequate sample was obtained from the biopsy
  * Clinical impression of malignant disease
Time from procedure to the initiation of treatment (in cases of malignancy) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifre L Maranki, M.D., Principal Investigator — Temple University

REFERENCES:
- [Background] Lee JG, Leung JW, Baillie J, Layfield LJ, Cotton PB. Benign, dysplastic, or malignant--making sense of endoscopic bile duct brush cytology: results in 149 consecutive patients. Am J Gastroenterol. 1995 May;90(5):722-6. PMID 7733076
- [Background] Glasbrenner B, Ardan M, Boeck W, Preclik G, Moller P, Adler G. Prospective evaluation of brush cytology of biliary strictures during endoscopic retrograde cholangiopancreatography. Endoscopy. 1999 Nov;31(9):712-7. doi: 10.1055/s-1999-73. PMID 10604612
- [Background] Kipp BR, Stadheim LM, Halling SA, Pochron NL, Harmsen S, Nagorney DM, Sebo TJ, Therneau TM, Gores GJ, de Groen PC, Baron TH, Levy MJ, Halling KC, Roberts LR. A comparison of routine cytology and fluorescence in situ hybridization for the detection of malignant bile duct strictures. Am J Gastroenterol. 2004 Sep;99(9):1675-81. doi: 10.1111/j.1572-0241.2004.30281.x. PMID 15330900
- [Background] Cote GA, Sherman S. Biliary stricture and negative cytology: what next? Clin Gastroenterol Hepatol. 2011 Sep;9(9):739-43. doi: 10.1016/j.cgh.2011.04.011. Epub 2011 Apr 22. No abstract available. PMID 21554986
- [Background] Draganov PV, Chauhan S, Wagh MS, Gupte AR, Lin T, Hou W, Forsmark CE. Diagnostic accuracy of conventional and cholangioscopy-guided sampling of indeterminate biliary lesions at the time of ERCP: a prospective, long-term follow-up study. Gastrointest Endosc. 2012 Feb;75(2):347-53. doi: 10.1016/j.gie.2011.09.020. PMID 22248602
- [Background] de Bellis M, Fogel EL, Sherman S, Watkins JL, Chappo J, Younger C, Cramer H, Lehman GA. Influence of stricture dilation and repeat brushing on the cancer detection rate of brush cytology in the evaluation of malignant biliary obstruction. Gastrointest Endosc. 2003 Aug;58(2):176-82. doi: 10.1067/mge.2003.345. PMID 12872082
- [Background] Fogel EL, deBellis M, McHenry L, Watkins JL, Chappo J, Cramer H, Schmidt S, Lazzell-Pannell L, Sherman S, Lehman GA. Effectiveness of a new long cytology brush in the evaluation of malignant biliary obstruction: a prospective study. Gastrointest Endosc. 2006 Jan;63(1):71-7. doi: 10.1016/j.gie.2005.08.039. PMID 16377319
- [Background] de Bellis M, Sherman S, Fogel EL, Cramer H, Chappo J, McHenry L Jr, Watkins JL, Lehman GA. Tissue sampling at ERCP in suspected malignant biliary strictures (Part 2). Gastrointest Endosc. 2002 Nov;56(5):720-30. doi: 10.1067/mge.2002.129219. No abstract available. PMID 12397282
- [Background] De Bellis M, Sherman S, Fogel EL, Cramer H, Chappo J, McHenry L Jr, Watkins JL, Lehman GA. Tissue sampling at ERCP in suspected malignant biliary strictures (Part 1). Gastrointest Endosc. 2002 Oct;56(4):552-61. doi: 10.1067/mge.2002.128132. No abstract available. PMID 12297773
- [Background] Weilert F, Bhat YM, Binmoeller KF, Kane S, Jaffee IM, Shaw RE, Cameron R, Hashimoto Y, Shah JN. EUS-FNA is superior to ERCP-based tissue sampling in suspected malignant biliary obstruction: results of a prospective, single-blind, comparative study. Gastrointest Endosc. 2014 Jul;80(1):97-104. doi: 10.1016/j.gie.2013.12.031. Epub 2014 Feb 19. PMID 24559784
- [Background] Chen YK, Pleskow DK. SpyGlass single-operator peroral cholangiopancreatoscopy system for the diagnosis and therapy of bile-duct disorders: a clinical feasibility study (with video). Gastrointest Endosc. 2007 May;65(6):832-41. doi: 10.1016/j.gie.2007.01.025. PMID 17466202
- [Background] Draganov PV, Lin T, Chauhan S, Wagh MS, Hou W, Forsmark CE. Prospective evaluation of the clinical utility of ERCP-guided cholangiopancreatoscopy with a new direct visualization system. Gastrointest Endosc. 2011 May;73(5):971-9. doi: 10.1016/j.gie.2011.01.003. Epub 2011 Mar 17. PMID 21419408
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Ramchandani M, Reddy DN, Gupta R, Lakhtakia S, Tandan M, Darisetty S, Sekaran A, Rao GV. Role of single-operator peroral cholangioscopy in the diagnosis of indeterminate biliary lesions: a single-center, prospective study. Gastrointest Endosc. 2011 Sep;74(3):511-9. doi: 10.1016/j.gie.2011.04.034. Epub 2011 Jul 7. PMID 21737076
- [Background] Siddiqui AA, Mehendiratta V, Jackson W, Loren DE, Kowalski TE, Eloubeidi MA. Identification of cholangiocarcinoma by using the Spyglass Spyscope system for peroral cholangioscopy and biopsy collection. Clin Gastroenterol Hepatol. 2012 May;10(5):466-71; quiz e48. doi: 10.1016/j.cgh.2011.12.021. Epub 2011 Dec 16. PMID 22178463